CLINICAL TRIAL: NCT01260441
Title: CPR Education of Patient Family Members Using CPR Anytime Training Program
Brief Title: An In-Hospital Family Member Cardiopulmonary Resuscitation (CPR) Education Program
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CRS-807120
Record Dates: First submitted 2010-11-29; First posted 2010-12-15 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Cardiac Arrest; Coronary Disease; Cardiovascular Risk Factors
MeSH Terms: conditions — Heart Arrest; Coronary Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard CPR (Active Comparator): Individuals will learn the Standard form of CPR (30:2, compressions:breathes) Main data points being collected over various increments are: 1) Comfort Level with using CPR 2) Secondary Training "multiplier effect" and 3) CPR Skills
  Interventions: Other: CPR Training using the Family and Friends CPR Anytime VSI Kit
- Chest Compressions Only CPR (Active Comparator): Individuals will learn the chest compression only form of CPR (no rescue breathes) Main data points being collected at various increments are: 1) Comfort Level with using CPR 2) Secondary Training "multiplier effect" and 3) CPR Skills
  Interventions: Other: CPR Training using the Family and Friends CPR Anytime VSI Kit

INTERVENTIONS:
Other: CPR Training using the Family and Friends CPR Anytime VSI Kit — Subjects will be trained using the American Heart Association's Family and Friends CPR Anytime Kit. Subjects will undergo training in-hospital and will be encouraged to take the kit home to share with their family members and friends.
  Other Names: Family and Friends CPR Anytime; American Heart Association Family and Friends CPR Anytime; CPR Anytime Video Self Instruction (VSI)

SUMMARY:
Each year in the United States, 300,000 people suffer from a Cardiac Arrest (CA), and of them, there is a 90% mortality rate. Out-of-Hospital arrests, in particular, have a 1-5% survival to hospital discharge. High quality CPR is crucial to lowering the mortality rate and increasing survival, yet only 15-30% of out-of-hospital CA victims receive bystander CPR. Studies have shown that prompt administration of CPR dramatically improves outcomes. In a recent study from Switzerland, lay bystander CPR doubled the survival rate at one month. Our study will look to train family members of at-risk cardiac patients in the skills of CPR through the American Heart Association's (AHA) CPR Anytime Friends and Family Personal Learning Program (CPR Anytime) to see if these family members are able to learn and perform quality CPR in the event that their family member should suffer a cardiac arrest.

DETAILED DESCRIPTION:
Using the AHA's CPR Anytime kit, we will work with family members of patients at high risk for a CA to learn lifesaving CPR skills. We will modify the AHA CPR video using the new AHA recommendations for bystanders which suggests doing chest compression only CPR. Using the original AHA video and our modified chest compression only video, we will randomize family members of patients at high risk for CA to one of these groups. Our research assistants will also be blinded to which video these subjects will be watching. After watching the video, we will have the subjects perform CPR on a mannequin using a CPR recording device that records chest compression rate and depth. We will follow up with the family members at 3 months, 6 months and 12 months to see if they retained their CPR knowledge and skills and to see if they had been in a situation where their CPR skills were needed and assess whether they performed their skills or not. We will also measure the number of people with whom the subjects shared their CPR Anytime kits-a quantity known as the multiplier effect to determine if they had shared the CPR Anytime kit with their family and friends, thereby increasing the possible number of lay persons trained in CPR and in turn able to perform bystander CPR if needed.

ELIGIBILITY:
Inclusion Criteria:

* Family member's of patients with known coronary disease or cardiovascular risk factors, such as history of diabetes and hypertension.

Exclusion Criteria:

* If someone is physically unable to undergo CPR Training
* Someone who has received CPR training in the past 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2007-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Subject Self-Confidence | within 30 minutes of CPR training
  We will administer a comprehensive post-training likert scale scoring survey to measure the subject's comfort level using their newly acquired CPR skills.
Secondary Training | 3 month increments over a 12 month period of time
  In addition, we will administer a telephone survey to measure the subject's secondary training through the CPR Anytime Kit.

SECONDARY OUTCOMES:
Assessing CPR Skills | 3 to 6 months post-training
  We will assess the subject's CPR skills by administering a 2-minute simulated CPR skills check recorded on a Laerdal Skillreporter ResusciAnne mannequin and video camera. The skills check will be conducted initially post training and at the 3-, 6-, and 12-month time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin S Abella, MD, MPhil, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Blewer AL, Leary M, Esposito EC, Gonzalez M, Riegel B, Bobrow BJ, Abella BS. Continuous chest compression cardiopulmonary resuscitation training promotes rescuer self-confidence and increased secondary training: a hospital-based randomized controlled trial*. Crit Care Med. 2012 Mar;40(3):787-92. doi: 10.1097/CCM.0b013e318236f2ca. PMID 22080629